CLINICAL TRIAL: NCT00709709
Title: Medical and Economic Medical Evaluation of Scan Multislice of Coronary Artery in Exploration of Stable Coronary Syndrome. Comparison With Quantitative Coronarography
Brief Title: Medical Evaluation of Scanner in Coronary Syndrome
Acronym: EVASCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P060105
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Syndrome
Keywords: stenosis; coronaropathy; stent; bypass surgery; suspect; known
MeSH Terms: conditions — Angina, Unstable; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Scan
  Interventions: Procedure: multislice coronary scan

INTERVENTIONS:
Procedure: multislice coronary scan — multislice coronary scan

SUMMARY:
Many recent publications have reported encouraging results on diagnostic cardiac multislice CT performance in 1) coronary artery disease, 2) coronary arterial bypass graft potency and 3) intrastent restenosis.

These single center studies were made on a limited number of patients (range, 50-130) and focused mainly on one of the indications mentioned above.

Moreover, results were often given after exclusion of low quality examinations. At last, no study has compared the diagnostic performance of the different CT systems '16, 40 and 64) in these populations.

DETAILED DESCRIPTION:
These single center studies were made on a limited number of patients (range, 50-130) and focused mainly on one of the indications mentioned above.

Moreover, results were often given after exclusion of low quality examinations. At last, no study has compared the diagnostic performance of the different CT systems '16, 40 and 64) in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients' ≥18 years, of both sexes
* Coronary angiography in patients with suspected of known CAD, instable clinical conditions.
* Clinical status allowing performance of coronary angiography 48 à 72h after CT examination
* Informed consent signed by patient

Exclusion Criteria:

* Patients in whom clinical status does not allow delayed coronary angiography
* Irregular heart rate, in particular atrial fibrillation
* Renal insufficiency (serum creatinine >150 µmol/l
* Radiology examination with use of iodin agent with 48h before) CT coronary
* K now intolerance to iodin agents
* Patients unable to hold breathing < 20 seconds
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Specificity and sensibility of scanner | visit 1

SECONDARY OUTCOMES:
Quality of coronary scanner imaging | visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Gueret, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France